CLINICAL TRIAL: NCT06578338
Title: A Study to Collect Data to Build Artificial INtelligence Derived Algorithms For Estimating Height and Weight in childRen (INFER)
Brief Title: Assessing a Height Artificial Intelligence Algorithm to Estimate Height of Children
Acronym: INFER
Status: Completed | Type: Observational
Sponsor: Danone Asia Pacific Holdings Pte, Ltd. (Industry)
Collaborators: KK Women's and Children's Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: SBB20R&31696-A
Record Dates: First submitted 2024-08-05; First posted 2024-08-29 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Growth; Stunting, Nutritional
Keywords: Growth; Height; Artificial Intelligence; Algorithm
MeSH Terms: conditions — Growth Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children aged above 24 months old and below 6 years of age: Children aged above 24 months old and below 6 years of age with no structural abnormalities of the lower limbs or orthopaedic conditions
  Interventions: Other: Physical height measurement

INTERVENTIONS:
Other: Physical height measurement — Physical height will be measured and images will be collected for AI to estimate the height

SUMMARY:
An exploratory study to explore the possibility of using computer vision algorithms to estimate a child's height using images taken by a healthcare professional or parents.

DETAILED DESCRIPTION:
This is an exploratory, observation, data-collection study that aims to evaluate the performance of a Height Artificial Intelligence (HAI) algorithm in a real world setting. Images will be collected by parents or healthcare professionals, together with physical height measurements. This data will be used to evaluate the accuracy of the algorithm and to explore potential improvements. Data on the acceptance and experience of using the algorithm will be collected for improvements.

ELIGIBILITY:
Inclusion Criteria:

* Children aged above 24 months old and below 6 years old.
* Parent(s) should have access to the internet and a smartphone or table to complete study questionnaires, take images and upload images.
* Parent(s) should be able to comprehend the content of the study and complete the study questionnaires in English.
* Written consent from parents and/or legally acceptable representative

Exclusion Criteria:

* Children who are unable to stand upright against a wall
* Children who are unable to cooperate with standing height measurement

Ages: 24 Months to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children aged above 24 months old and below 6 years of age with no physical deformities
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2024-09-09 (Actual); Primary Completion 2025-03-04 (Actual); Study Completion 2025-03-04 (Actual)

PRIMARY OUTCOMES:
Accuracy of the height AI (cm) | 2 days
  Accuracy of the Height AI (cm) in a clinic and in a home setting, derived from:
  1. The height AI prediction from images collected
  2. The physical height measurements of subjects using WHO standard height measurement

SECONDARY OUTCOMES:
Accuracy of the Weight AI (kg) | 2 days
  Accuracy of the Weight AI (kg) in a clinic and in a home setting, derived from:
  1. The weight prediction from the standing images collected in this study
  2. The WHO standard weight measurement of subjects

OTHER OUTCOMES:
Assessments by the parent on usability of the AI in a home-setting via study questionnaire | 2 days
  1. Ease of collecting images (very easy to very difficult)
  2. Acceptable range of height & weight difference between AI prediction & WHO measurement (between ≤1cm and >5cm)
  3. Frequency of measuring child's height & weight at home (never,< 1/month, at least <1/month, at least 1 per 2 weeks,at least 1/week,> 1/week,daily)
  4. Usefulness of using digital tool to measure child's height & weight at home (Very useful to Not very useful)
  5. Frequency of using digital tool to measure child's height & weight at home (never,<1/month, at least 1/month, at least 1 per 2 weeks,at least 1/week,>1/week,daily)
  6. Likelihood and reason of using a digital tool to measure child's height & weight at home (Very Likely to Very unlikely)
  7. Sharing the child's height & weight measured using digital tool with others (Very Likely to Very unlikely)
  8. Use of mobile apps to track child's height & weight (free text)
  9. Other features/tools useful to measure child's height & weight (free text)
Assessments by the investigator on usability of the AI in a clinic-setting via a questionnaire | 2 days
  1. Acceptable range of height and weight difference between the height and weight AI from the WHO measurement (≤ 1cm, ≤ 2cm, ≤ 3cm, ≤ 4cm, ≤5cm, >5cm)
  2. Likelihood of using a digital tool to measure a child's height and weight in a clinical setting (Very Likely, Likely, Neutral, Unlikely, Very unlikely)
  3. Likelihood of recommending parents to use a digital tool to measure their child's height and weight in a clinical setting (Very Likely, Likely, Neutral, Unlikely, Very unlikely)
  4. Other features/tools they find useful to measure the child's height and weight (free text)
Assessments by the investigator on ease of collecting images in a clinic-setting via a questionnaire | 2 days
  Investigator's assessment on the ease of collecting the images [Very Easy, Easy, Normal, Difficult, Very Difficult]

CONTACTS AND LOCATIONS:
Overall Officials: Fabian Yap, MBBS, Principal Investigator — KK Women's and Children's Hospital
Locations (1):
- KK Women's and Children's Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yap F, Lee YS, Aw MMH. Growth Assessment and Monitoring during Childhood. Ann Acad Med Singap. 2018 Apr;47(4):149-155. PMID 29777245
- [Background] Schmidhuber J. Deep learning in neural networks: an overview. Neural Netw. 2015 Jan;61:85-117. doi: 10.1016/j.neunet.2014.09.003. Epub 2014 Oct 13. PMID 25462637